CLINICAL TRIAL: NCT03165409
Title: Economic Burden of Adverse Events Associated With Follow-Up Frequency Among Patients With Metastatic Melanoma
Brief Title: Cost of Adverse Events Related to How Often Follow-Up Occurs Among Patients With Cancer That Has Spread
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-789
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Nivolumab — Melanoma intervention
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab — Melanoma intervention
  Other Names: BMS-734016; Yervoy

SUMMARY:
This study is a real-world retrospective claims analysis to assess and compare AE-related HCRU and medical costs among patients with different follow-up frequency after initiating a melanoma therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metastatic melanoma
* Initiated at least 1 treatment for metastatic melanoma after 2011
* Continuous enrollment in their healthcare plan for at least 6 months before and at least 6 weeks after the index date
* Patients who received at least 1 dose of study drug in CA209-067

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who were diagnosed with metastatic melanoma and initiated at least 1 treatment for metastatic melanoma after 2011 will be identified from the IMS PharMetrics Plus US Claims Database and included in the study sample. Patients must have had continuous enrollment in their healthcare plan for at least 6 months before and at least 6 weeks after the index date. The population from the CheckMate-067 (CA209-067) clinical trial will also be included. The population consists of all patients who received at least 1 dose of study drug.
Sampling Method: Non-Probability Sample
Enrollment: 1828 (Actual)
Dates: Start 2017-02-27 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Composite monthly incidence rate of adverse events (AEs), AE-related healthcare resource utilization, and medical costs among the metastatic melanoma patients with less frequent general outpatient visits | Approximately 5 years
Composite monthly incidence rate of adverse events (AEs), AE-related healthcare resource utilization, and medical costs among the metastatic melanoma patients with more frequent general outpatient visits | Approximately 5 years
Treatment-related and all-cause AE costs for nivolumab/ipilimumab combination therapy for metastatic melanoma | Approximately 5 years
Treatment-related and all-cause AE costs for nivolumab monotherapy for metastatic melanoma | Approximately 5 years
Treatment-related and all-cause AE costs for ipilimumab monotherapy for metastatic melanoma | Approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Bristol-Myers Squibb, Princeton, New Jersey, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx